CLINICAL TRIAL: NCT04603911
Title: An Investigator-Initiated, Double-Blind, Patient-Controlled, Randomized Control Trial Comparing the Effectiveness of Liposomal Bupivacaine to a Solution of Bupivacaine, Epinephrine Clonidine and Dexamethasone in Bilateral, Single Shot, Erector Spinae Plane Blocks During Oncoplastic Breast Surgery
Brief Title: RCT Comparing ESPB Solutions in Breast Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00000228
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: bilateral breast surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Epinephrine; Dexamethasone; Clonidine; Reference Standards

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Control arm will receive standard of care solution for the ESPB block
  Interventions: Drug: Bupivacaine, epinephrine, dexamethasone, and clonidine
- Liposomal Bupivicaine (Active Comparator): Liposomal Bupivicaine arm will receive Liposomal Bupivicaine for the ESPB block
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — The liposomal bupivacaine used in the research study has been approved by the U.S. Food and Drug Administration (FDA) for use in humans for pain management. The specific approved uses are postsurgical single-dose wound infiltration analgesia and brachial plexus nerve block. In this study, we will be using liposomal bupivacaine in an additional way by infiltrating liposomal bupivacaine in a tissue plane to numb the nerves that provide sensation over the chest.
  Other Names: Exparel
  Arms: Liposomal Bupivicaine
Drug: Bupivacaine, epinephrine, dexamethasone, and clonidine — The medications that are typically administered as a solution in this block include bupivacaine, epinephrine, dexamethasone, and clonidine.
  Other Names: Standard Preparation
  Arms: Control

SUMMARY:
The object of our research is to investigate the relative efficacy of liposomal bupivacaine administered via an Erector Spinae Plane (ESP) block as compared to our standard of care medication solution of (bupivacaine mixed with epinephrine, dexamethasone, and clonidine) for pain management in subjects undergoing bilateral surgical intervention for breast cancer. This will be an investigator-initiated, double-blind, patient-controlled, randomized control trial comparing pain scores at 48 hours after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 75 years of age at screening
2. Scheduled to undergo oncoplastic bilateral mastectomy and reconstruction surgery at Tufts Medical Center

Exclusion Criteria:

1. Adults unable to consent (inability to read, write, or has some impairment that hampers consent process or documentation, or cognitively impaired adults)
2. Pregnant women
3. Pregnant minors
4. Woman of childbearing potential who are unwilling or unable to complete a pregnancy test
5. Minors i.e., individuals who are not yet adults (neonates, children, teenagers)
6. Wards of the state
7. Non-viable neonates
8. Neonates of uncertain viability
9. Prisoners
10. Adults with known allergy, hypersensitivity, intolerance or contraindication to study medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Pain Score at 48 hours | 48 hours
  Pain score will be recorded using a visual analogue scale (VAS) where 0 is no pain and 10 is unbearable pain.
  Pain will be recorded for the right and left side independently.

SECONDARY OUTCOMES:
Pain Scores at 6, 12, 18, 24, 30, 38, 42, and 72 hours | 72 hours
  Pain score will be recorded using a visual analogue scale (VAS) where 0 is no pain and 10 is unbearable pain.
  Pain will be recorded for the right and left side independently.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States